CLINICAL TRIAL: NCT02098538
Title: A Phase II Study of Regorafenib in Patients With Progressive, Recurrent/Metastatic Adenoid Cystic Carcinoma
Brief Title: Regorafenib in Patients With Progressive, Recurrent/Metastatic Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-244
Record Dates: First submitted 2014-03-24; First posted 2014-03-28 (Estimated); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-11

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Regorafenib; 13-244
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — regorafenib

ARMS (1):
- patients with adenoid cystic carcinoma (Experimental): This is a single-arm phase II study of patients with progressive, recurrent/metastatic adenoid cystic carcinoma (R/M ACC) treated with regorafenib.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — All eligible patients will receive a starting regorafenib dose of 120 mg daily taken orally for 3 weeks in a 4-week cycle. Patients for whom regorafenib dose reduction was not performed or required may have their treatment dose increased to the FDA-approved dose of 160 mg daily orally for 3 weeks in a 4-week cycle in cycle #2 or beyond (this is not mandatory). RECIST v1.1 tumor assessments will be made at baseline (CT or MRI) and then approximately every 2 cycles (or every 8 weeks (+/- 1 week)). After 10 months, imaging will be done every 3 cycles (or every 12 weeks (+/- 1 week)). Patients may remain on study until progression of disease or unacceptable toxicity

SUMMARY:
Regorafenib is an oral medication that can interfere with cancer cell growth and reduce the growth of blood vessels around tumors. This study will help find out if regorafenib is a useful drug for treating patients with adenoid cystic carcinomas. Regorafenib has been approved by the Food and Drug Administration (FDA) for use in other cancers, but remains an experimental drug that has not yet been approved for use in adenoid cystic carcinoma.

In this study, the patient will initially be treated with a dose of regorafenib that is lower than what the FDA approved for other cancers in an attempt to decrease the risk of side effects. It is possible that this lower starting dose may not be as effective as the higher FDA approved dose. If the patient does well with the lower dose for at least a month on treatment, the physician may consider increasing the dose to the FDA approved dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically confirmed adenoid cystic carcinoma. Cancers arising from non-salivary gland primary sites are allowed.
* Patients must have recurrent and/or metastatic disease not amenable to potentially curative surgery or radiotherapy.
* At least 2 weeks must have elapsed since the end of prior systemic treatment (4 weeks for bevacizumab- containing regimens) or radiotherapy with resolution of all treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia, lymphopenia, or hypothyroidism). Any number of prior therapies for recurrent/metastatic ACC are allowed.
* Patients must have RECIST v1.1 measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan.
* Patients must have documentation of a new or progressive lesion on a radiologic imaging study performed within 6 months prior to study enrollment (progression of disease over any interval is allowed) and/or new/worsening disease related symptoms within 6 months prior to study enrollment. Note: This assessment will be performed by the treating investigator. Evidence of progression by RECIST criteria is not required.
* Patients must have archival tissue from the primary tumor or metastases available for correlative studies. Either a paraffin block or twenty unstained slides are acceptable. If twenty slides are not available, a lesser amount may be acceptable after discussion with the Principal Investigator, Dr. Alan L. Ho.
* Patients must agree to undergo biopsy of a malignant lesion. Biopsies do not need to be done if either the investigator or person performing the biopsy judges that no tumor is accessible for biopsy or that biopsy poses too great of a risk to the patient. Patients may also be exempt if frozen tumor tissue has been collected within 12 months of study enrollment that the Principal Investigator deems is appropriate/sufficient for analysis on this protocol.
* Age ≥ 18 years.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%,).
* Life expectancy of at least 12 weeks (3 months) as determined by the investigator.
* Life expectancy of at least 12 weeks (3 months) as determined by the investigator.
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

  * Total bilirubin ≤ 1.5 x the upper limits of normal (ULN) Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Lipase ≤ 1.5 x the ULN
  * Amylase ≤ 1.5 x the ULN Serum creatinine ≤ 1.5 x the ULN or calculated creatinine clearance >60 ml/min
  * Platelet count ≥ 100,000 /mm3, hemoglobin (Hb) ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm3. Blood transfusion to meet the inclusion criteria will not be allowed.
* Women of childbearing potential must have a negative serum pregnancy test performed within 2 weeks prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the consent form until at least 3 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* Concurrent anti-cancer therapy (chemotherapy, definitive radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment. Concurrent therapy with bisphosphonates or denosumab for bone metastases is allowed.

Palliative radiation to non-target lesions is also allowed.

* Prior use of regorafenib.
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management.
* Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form).
* Concurrent use of strong CYP3A4 inhibitors (e.g. clarithromycin, grapefruit juice, itraconazole, ketoconazole, nefazodone, posaconazole, telithromycin, and voriconazole). or strong CYP3A4 inducers (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort).
* Use of any herbal remedy (e.g. St. John's wort [Hypericum perforatum])
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Active or clinically significant cardiac disease including:

Congestive heart failure - New York Heart Association (NYHA) > Class II.

* Active coronary artery disease that is not medically treated.
* Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
* Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.

  * Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin) is not allowed if the medication dose and/or INR/PTT are not considered stable by the treating physician. If the dose and/or INR/PTT are stable, therapeutic anticoagulation with Vitamin-K antagonists is allowed with close monitoring. Anticoagulation with heparin or heparinoids is allowed.
  * Evidence or history of bleeding diathesis or coagulopathy.
  * Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
  * Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment.
  * Subjects with a past or current diagnosis of another malignancy that will interfere with conduct of the trial. Patients with past or current cancer diagnoses other than ACC are allowed to enroll if the investigator believes it will not interfere with trial conduct.
  * Patients with phaeochromocytoma.
  * Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
  * Active infection that would impair the ability of the patient to receive study treatment.
  * Symptomatic metastatic brain or leptomeningeal tumors (asymptomatic or treated metastatic brain and leptomeningeal tumors are allowed).
  * Presence of a non-healing wound or non-healing ulcer that is not tumor related.
  * Renal failure requiring hemo-or peritoneal dialysis.
  * Patients with seizure disorder requiring medication.
  * Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
  * History of organ allograft (including corneal transplant).
  * Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
  * Any malabsorption condition.
  * Women who are pregnant or breast-feeding.
  * Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
  * Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Adenoid Cystic Carcinoma
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Adenoid Cystic Carcinoma
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive With and Without Disease Progression
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Adenoid Cystic Carcinoma
Number analyzed (Participants) | 38
Participants
  Participants alive without disease progression | 4
  Participants alive with disease progression | 6
  Not evaluable | 28

2. Primary Outcome: Best Overall Response Rate
Description: (BOR = CR+PR) documented by RECIST v1.1 criteria
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Adenoid Cystic Carcinoma
Number analyzed (Participants) | 38
Participants
  Participants with CR+PR | 1
  Participants without CR+PR | 37

3. Secondary Outcome: Number of Participants Evaluated for Adverse Events
Description: Safety will be assessed in terms of AEs, laboratory data and vital sign data, which will be collected for all patients. Appropriate summaries of these data will be presented. AE will be listed individually per patient according to CTCAE version 4.0, and the number of patients experiencing each AE will be summarized. The safety population will comprise all patients who receive at least one dose of study treatment.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Adenoid Cystic Carcinoma
Number analyzed (Participants) | 38
Participants | 38

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patients With Adenoid Cystic Carcinoma
All-Cause Mortality (participants affected / at risk) | 28/38
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Adenoid Cystic Carcinoma (N=38)
Abdominal Pain (Gastrointestinal disorders) | 2
Alanine aminotransferase, increased (Investigations) | 2
Aspartate aminotransferase, increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bilirubin, increased (Hepatobiliary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 1
Lymphocyte count, decreased (Investigations) | 4
Lethargy (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1
Platelet count, decreased (Blood and lymphatic system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 5
Soft tissue infection (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Adenoid Cystic Carcinoma (N=38)
Alanine aminotransferase, increased (Investigations) | 27
Aspartate aminotransferase, increased (Investigations) | 29
Alopecia (Skin and subcutaneous tissue disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Alkaline phosphatase, increased (Investigations) | 25
Anorexia (Metabolism and nutrition disorders) | 13
Anal ulcer (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 2
Anemia (Blood and lymphatic system disorders) | 18
Abdominal pain (Gastrointestinal disorders) | 9
Activated partial thromboplastin time prolonged (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Blurred vision (Eye disorders) | 9
Bilirubin, increased (Investigations) | 28
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Burn (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Cataract (Eye disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Constipation (Gastrointestinal disorders) | 15
Chills (General disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Cholesterol high (Investigations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Creatinine increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 16
Dry skin (Skin and subcutaneous tissue disorders) | 8
Dry eye (Eye disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Depression (Psychiatric disorders) | 2
Dry mouth (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
External ear pain (Ear and labyrinth disorders) | 1
Eye infection (Infections and infestations) | 1
Edema limbs (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Facial nerve disorder (Nervous system disorders) | 2
Facial pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fever (General disorders) | 8
Floaters (Eye disorders) | 3
Fatigue (General disorders) | 32
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Hemoglobin, increased (Investigations) | 8
Headache (Nervous system disorders) | 11
Hearing impaired (Ear and labyrinth disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 17
Hypophosphatemia (Metabolism and nutrition disorders) | 22
Hypertension (Vascular disorders) | 30
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 27
Hyperglycemia (Metabolism and nutrition disorders) | 37
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypothyroidism (Endocrine disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 14
Insomnia (Psychiatric disorders) | 3
Irregular menstruation (Reproductive system and breast disorders) | 1
Lipase increased (Investigations) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count, decreased (Investigations) | 13
Lip pain (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal & conn tissue disorder, other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Malaise (General disorders) | 2
Mucositis, oral (Gastrointestinal disorders) | 6
Mucosal infection (Infections and infestations) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 15
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuralgia (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Non-cardiac chest pain (General disorders) | 1
Oral cavity fistula (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 6
Oral pain (Gastrointestinal disorders) | 17
Oral dysesthesia (Gastrointestinal disorders) | 3
Otitis media (Infections and infestations) | 1
Pain (General disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Platelet count, decreased (Blood and lymphatic system disorders) | 20
Pruritus (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 28
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 15
Pericarditis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Periorbital edema (Eye disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Paresthesia (Nervous system disorders) | 6
Rash, acneiform (Skin and subcutaneous tissue disorders) | 2
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 17
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Sinus tachycardia (Cardiac disorders) | 6
Sinusitis (Infections and infestations) | 2
Serum amylase increased (Investigations) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 10
Tooth infection (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary frequency (Renal and urinary disorders) | 7
Urinary tract infection (Infections and infestations) | 1
Urinary tract pain (Renal and urinary disorders) | 2
Vascular disorders, other (Vascular disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Investigations) | 15
White blood cell, decreased (Blood and lymphatic system disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT02098538/Prot_SAP_000.pdf